CLINICAL TRIAL: NCT05377931
Title: Ocular and Cardiac Effects of Mobile Battle Ground Games
Brief Title: Ocular and Cardiac Effects of Battle Ground
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Lecturer of Ophthalmology, Benha University
Other Study IDs: RC 10-22
Record Dates: First submitted 2022-05-12; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: COVID-19; Accommodation Spasm; Tachycardia; Stress Reaction; Cardiac Arrhythmia
Keywords: Battle ground games; Accommodation; Spasm; Eye strain; Pulse disorder; Tachycardia
MeSH Terms: conditions — COVID-19; Spasm; Tachycardia; Fractures, Stress; Arrhythmias, Cardiac; Asthenopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal subjects users of battle ground games (Group 1): Subjects with no history of any medical diseases that are using mobile battle ground games for average 2 hours per day.
  Interventions: Diagnostic Test: Changes in heart pulse rate; Diagnostic Test: Changes in eye strain
- Post COVID-19 users of battle ground games (Group 2): Adults with a recent history of COVID-19 (average of 6 months after onset of the disease) that returned to their normal life style and are using mobile battle ground games.
  Interventions: Diagnostic Test: Changes in heart pulse rate; Diagnostic Test: Changes in eye strain
- Normal subjects not playing mobile games (Groups 3): Normal subjects that are not using any action mobile games.
  Interventions: Diagnostic Test: Changes in heart pulse rate; Diagnostic Test: Changes in eye strain

INTERVENTIONS:
Diagnostic Test: Changes in heart pulse rate — Measuring heart pulse rate using a wrest smart watch.
  Other Names: Pulse oximeter changes
Diagnostic Test: Changes in eye strain — Changes in Accommodation measured by auto refractometer before and after mobile battle ground gaming.

SUMMARY:
Mobile battle ground games are widely used in various age groups, there are ocular and cardiac affection that may affect users of this type of action games.

DETAILED DESCRIPTION:
The aim of this study is to assess the possible ocular and cardiac changes that may affect users of this type of mobile games in real life among various age groups and especially in adults with history of recent corona virus (COVID-19) disease. There is no medical recommendations about the time and the hazards of using this games for longer periods in real practice.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects that are playing or not playing action mobile battle ground games will be included.
* Post COVID-19 subjects with average 6 months of infection and are playing mobile battle. Ground games will be included.

Exclusion Criteria:

* Subjects that refuse to enter the study.
* Users of mobile battle ground games with other diseases that may affect ocular and cardiac assessment as diabetic eye disease, cardiac congenital anomalies or recent cardiac or ocular surgery.

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Subjects that are using action mobile games during their leisure and are members of faculty of medicine, Banha university and are seeking to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-02-10 (Estimated); Study Completion 2023-02-20 (Estimated)

PRIMARY OUTCOMES:
Changes in heart pulse rate | During playing mobile battle ground games
  Changes in pulse in each group members measured by smart wrest watch in pulse beat/per minute.

SECONDARY OUTCOMES:
Changes in accommodation | Before and immediately after mobile battle ground games
  Changes in eye accommodation measured by auto refractometer in diopter (D).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Abdelshafy, MD, Study Chair — Benha University
Locations (1):
- Ahmed Abdelshafy, Banhā, QA, Egypt

IPD SHARING:
Plan to Share IPD: Undecided